CLINICAL TRIAL: NCT06136182
Title: Clinical Outcome of Pericardial Closure Using Gentrix Following Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 016.SUR.2023.M
Record Dates: First submitted 2023-07-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Clinical Outcome of Pericardial Closure Using Gentrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pericardial Closure Using Gentrix Following Cardiac Surgery — To determine feasibility and effectiveness of Gentrix for cardiac use, and if this product is patient population specific.

SUMMARY:
A descriptive comparative project will be conducted to determine if there is a difference in outcomes for adult patients requiring pericardial reconstruction using CorMatrix compared to Gentrix

DETAILED DESCRIPTION:
A descriptive, comparative project will be conducted utilizing a retrospective chart review on patients at Methodist Mansfield Medical Center(MMMC) undergoing cardiac surgery requiring pericardial repair between the dates of January 1, 2017 through December 31, 2022. The project will compare outcomes of a pre- and post-intervention following use of Gentrix ECM and the CorMatrix Extracellular Matrix(ECM) pericardial patch using information gathered from the patient's electronic health record (EHR). The main outcome measures of post-operative Length of Stay(LOS), all-cause unplanned readmission within 30 days, and significant pleural effusion requiring thoracentesis within 30-days and 60 days as well as long-term (12 months) patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Must have undergone a Coronary Artery Bypass Grafting(CABG) or valve repair/replacement surgery requiring pericardial reconstruction.

CABG or valve repair/replacement surgery must have been either elective or urgent status

Exclusion Criteria:

-CABG or valve repair/replacement surgery classified as emergent status Surgery classified as redo-sternotomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Must have undergone a CABG or valve repair/replacement surgery requiring pericardial reconstruction.
  * CABG or valve repair/replacement surgery must have been either elective or urgent status
Sampling Method: Probability Sample
Enrollment: 489 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-05-12 (Estimated); Study Completion 2024-05-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative hospital LOS | 30 days
  30-day all-cause unplanned readmissions after discharge
  * Significant pleural effusion requiring thoracentesis within 30 days of surgery
  * Significant pleural effusion requiring thoracentesis within 60 days of surgery

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Research Institute at Methodist Health System, Dallas, Texas
  - Methodist Dallas Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data Might be available by 2024 for up to 4 years
Access Criteria: All study-related documents will be retained by the clinical research institute (CRI) until at least three years after study completion or according to local laws, whichever is longer

REFERENCES:
- [Background] Bachar, B and Manna, B. (2022, August 8). Coronary Artery Bypass Graft. National Library of Medicine. https://www.ncbi.nlm.nih.gov/books/NBK507836/
- [Background] Rego A, Cheung PC, Harris WJ, Brady KM, Newman J, Still R. Pericardial closure with extracellular matrix scaffold following cardiac surgery associated with a reduction of postoperative complications and 30-day hospital readmissions. J Cardiothorac Surg. 2019 Mar 15;14(1):61. doi: 10.1186/s13019-019-0871-5. PMID 30876459
- [Background] Valve repair or replacement (2022). In The Texas Heart Institute. https://www.texasheart.org/heart-health/heart-information-center/topics/valve-repair-or-replacement/